CLINICAL TRIAL: NCT00430898
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of the Safety, Efficacy, and Pharmacokinetics of Multiple Doses of Basiliximab, With Concomitant Corticosteroids, in Steroid-Refractory Ulcerative Colitis
Brief Title: Basiliximab in Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerimon Pharmaceuticals (Industry)
Responsible Party: Cerimon Pharmaceuticals, Inc, Cerimon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSX-001
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis basiliximab
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Basiliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Placebo (Placebo Comparator): Placebo to mimic 40 mg of Simulect
  Interventions: Drug: Basiliximab
- 2. 40 mg Simulect (Experimental): 40 mg of Simulect
  Interventions: Drug: Basiliximab

INTERVENTIONS:
Drug: Basiliximab — 3 doses of 40mg, IV at baseline, week 2, and week 4
  Other Names: Simulect

SUMMARY:
The purpose of this study is to assess the safety, effectiveness and pharmacokinetics of two levels of intravenous basiliximab in ulcerative colitis, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

In addition to others,

* Men or women age 18-75
* Diagnosis of ulcerative colitis confirmed through screening endoscopy.
* Extent of disease must involve at least the left colon
* Moderate to severe disease (Mayo Score 6-12). Systemic features of tachycardia, fever, and/or significant anemia should not be present.
* Inadequate response despite treatment with prednisone 40 - 50 mg/day (or other oral steroid at equivalent dose) orally for a minimum of 14 days immediately preceding study entry

Exclusion Criteria:

In addition to other protocol-defined conditions,

* Pregnancy
* Stool study that shows presence of ova and parasites, significant bacterial pathogens, or C. difficile toxin
* Colitis that is indeterminate, suggestive of Crohn's disease, or isolated to the rectum, based on endoscopic and/or biopsy findings
* Severely ill patients as evidenced by protocol-defined systemic criteria
* Chest radiograph abnormalities consistent with an infectious process
* History of colonic dysplasia
* HIV infection
* Known viral Hepatitis B or C infection
* History of or exposure to tuberculosis within 6 months before study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in Mayo Score, Safety | At week 8

SECONDARY OUTCOMES:
Clinical remission at week 4; clinical response at weeks 4 and 8; use of rescue medication; hospitalization or colectomy; and concomitant steroid use | at week 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Levitt, MD, PhD, Study Director — Cerimon Pharmaceuticals
Locations (61):
- United States (25):
  - Anaheim, California
  - Roseville, California
  - Golden, Colorado
  - Littleton, Colorado
  - Hollywood, Florida
  - Jacksonville, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Urbana, Illinois
  - Indianapolis, Indiana
  - Topeka, Kansas
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Troy, Michigan
  - Egg Harbor Twp, New Jersey
  - Great Neck, New York
  - New York, New York
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Sewickley, Pennsylvania
  - Germantown, Tennessee
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
- Leuven, Belgium
- Czechia (4):
  - Mladá Boleslav
  - Prague
  - Tábor
  - Ústí nad Orlicí
- India (9):
  - Bangalore
  - Hyderabaad
  - Kochi
  - Kolkata
  - Lucknow
  - Ludhiana
  - Mumbai
  - New Delhi
  - Visakhapatnam
- Poland (6):
  - Gdansk
  - Krakow
  - Poznan
  - Sopot
  - Warsaw
  - Wroclaw
- Russia (3):
  - Moscow
  - Samara
  - Smolensk
- Slovakia (4):
  - Bratislava
  - Nitra
  - Nové Mesto nad Váhom
  - Prešov
- Ukraine (4):
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
- United Kingdom (5):
  - Bristol
  - Derbyshire
  - London
  - Stoke-on-Trent
  - Wigan

REFERENCES:
- [Derived] Sands BE, Sandborn WJ, Creed TJ, Dayan CM, Dhanda AD, Van Assche GA, Gregus M, Sood A, Choudhuri G, Stempien MJ, Levitt D, Probert CS. Basiliximab does not increase efficacy of corticosteroids in patients with steroid-refractory ulcerative colitis. Gastroenterology. 2012 Aug;143(2):356-64.e1. doi: 10.1053/j.gastro.2012.04.043. Epub 2012 Apr 28. PMID 22549092